CLINICAL TRIAL: NCT01738022
Title: Mechanisms of Pharyngeal Collapse in Sleep Apnea, Study C
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012P000957C; 1R01HL102321-01A1 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-30 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Pathophysiology
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — heliox; Sulfur Hexafluoride; Neon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gas mixture administration (Experimental): Subjects will breathe different gas mixtures with different densities and viscosity for brief periods in order to promote changes in peak inspiratory flow
  Interventions: Other: Administration of gas mixtures

INTERVENTIONS:
Other: Administration of gas mixtures
  Other Names: Heliox; Sulfur-hexafluoride; Neon

SUMMARY:
In obstructive sleep apnea (OSA), the upper airway recurrently closes during sleep. The mechanisms that lead to airway closure are not completely understood. Models to study mechanisms of airway collapse have been proposed. However, these models have not been tested in the human upper airway. Gas density and viscosity are different gas properties that influence upper airway collapse and are variables of different models. In this study, subjects will breathe gas mixtures of different densities and viscosities for brief periods of time in order to test those models.

DETAILED DESCRIPTION:
Models to study mechanisms of airway collapse have been proposed. However, these models have not been tested in the human upper airway. Gas density and viscosity are different gas properties that influence upper airway collapse and are variables of different models.

In this study, subjects will breathe gas mixtures of different densities (helium and sulfur-hexafluoride) or viscosity (neon) for brief periods of time during flow-limited breaths. Flow limitation will be induced by sustained reductions of continuous positive airway pressure (CPAP). The investigators will test some models of upper airway collapse by observing if flow while breathing different gas mixtures scales according to the differences in density and viscosity.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects or patients with OSA

Exclusion Criteria:

* Any unstable cardiac condition (other than well controlled hypertension) or pulmonary problems.
* Any medication known to influence breathing, sleep/arousal or muscle physiology
* Concurrent sleep disorders (insomnia, narcolepsy, central sleep apnea or parasomnia)
* Claustrophobia
* Inability to sleep supine
* Allergy to lidocaine or oxymetazoline hydrochloride
* For women: Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12-08 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Difference in peak inspiratory flow | 10 - 15 seconds
  Observed peak inspiratory flow while breathing different gas mixtures will be compared to model predicted flows.
  Subjects will breathe different gas mixtures for 2 consecutive breaths only. Therefore the time frame is equal to one breath before gas mixture administration and two breaths after (usually 10-15 seconds).

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States